CLINICAL TRIAL: NCT05614245
Title: A Phase 1, Open-Label, Adjuvant Dose-Escalation, Randomized Study to Evaluate the Safety and Immunogenicity of VBI-2901e, a Trivalent Coronavirus Vaccine Candidate Adjuvanted With Aluminum Phosphate and E6020 in Healthy Adults Previously Vaccinated With Licensed COVID-19 Vaccines
Brief Title: Safety, Tolerability, and Immunogenicity of Trivalent Coronavirus Vaccine Candidate VBI-2901e With E6020 Adjuvant
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was halted prematurely prior to enrollment of first participant based on study sponsor's decision to prioritize clinical development of VBI-2901a.
Sponsor: VBI Vaccines Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VBI-2901e-CT01
Record Dates: First submitted 2022-11-02; First posted 2022-11-14 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Coronavirus Infections
Keywords: COVID-19; SARS-CoV-2; SARS-CoV-1; MERS-CoV; vaccine; enveloped virus-like particle (eVLP); coronavirus; adjuvant; E6020
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group G1, Subgroup G1-A (Experimental): 10 participants aged 18-40 years to receive one dose of VBI-2901e at 5 µg spike protein and 1 µg E6020 per dose at Day 1
  Interventions: Biological: VBI-2901e
- Group G1, Subgroup G1-B (Experimental): 10 participants aged 18-40 years to receive two doses of VBI-901e at 5 µg spike protein and 1 µg E6020 per dose at Day 1 and Day 28
  Interventions: Biological: VBI-2901e
- Group G2, Subgroup G2-A (Experimental): 10 participants aged 18-40 years to receive one dose of VBI-2901e at 5 µg spike protein and 3 µg E6020 per dose at Day 1
  Interventions: Biological: VBI-2901e
- Group G2, Subgroup G2-B (Experimental): 10 participants aged 18-40 years to receive two doses of VBI-901e at 5 µg spike protein and 3 µg E6020 per dose at Day 1 and Day 28
  Interventions: Biological: VBI-2901e
- Group G3, Subgroup G3-A (Experimental): 10 participants aged 18-40 years to receive one dose of VBI-2901e at 5 µg spike protein and 10 µg E6020 per dose at Day 1
  Interventions: Biological: VBI-2901e
- Group G3, Subgroup G3-B (Experimental): 10 participants aged 18-40 years to receive two doses of VBI-901e at 5 µg spike protein and 10 µg E6020 per dose at Day 1 and Day 28
  Interventions: Biological: VBI-2901e

INTERVENTIONS:
Biological: VBI-2901e — Intramuscular injection of VBI-2901e, an investigational trivalent coronavirus vaccine that contains three coronavirus spike proteins with aluminum phosphate and E6020 adjuvants

SUMMARY:
VBI-2901e is an investigational vaccine candidate that uses enveloped virus-like particles (eVLPs) to express the spike proteins of three coronaviruses: SARS-CoV-2 (the virus that causes COVID-19 disease), SARS-CoV-1 and MERS-CoV. The trivalent vaccine candidate is designed to induce neutralizing antibody and cell-mediated immune responses against the spike protein of the original strain of SARS-CoV-2 coronavirus, variants and subvariants of SARS-CoV-2 (such as Beta, Delta and Omicron BA.5) and other related coronaviruses that could emerge in the future. VBI-2901e contains two adjuvants: aluminum phosphate and E6020. The role of the adjuvants is to create a stronger immune response to the vaccine.

This Phase 1 study will be an open-label study of VBI-2901e comparing three dose levels of the E6020 adjuvant component (1, 3, or 10 µg per dose) in adults 18 to 40 years of age who had previously received two or more vaccinations with licensed COVID-19 vaccine(s). VBI-2901e at each dose level of E6020 will be administered as either a single dose or two-dose regimen. The purpose of the study is to test the safety of VBI-2901e and to learn more about its ability to boost immune responses against SARS-CoV-2 and the two related coronaviruses SARS-CoV-1 and MERS-CoV.

DETAILED DESCRIPTION:
VBI-2901e is an investigational trivalent COVID-19 vaccine candidate that comprises enveloped virus-like particles (eVLPs) expressing the spike proteins of the betacoronaviruses SARS-CoV-2, SARS-CoV-1 and MERS-CoV and the adjuvants aluminum phosphate and E6020 (a toll-like receptor 4 agonist). The study will enroll participants 18 to 40 years of age who have previously received two or more vaccinations with licensed COVID-19 vaccine(s) and will test one or two intramuscular doses of VBI-2901e containing 5 μg of SARS-CoV-2 spike protein, 165 µg of aluminum phosphate and 1, 3 or 10 µg of E6020. VBI-2901e is designed to induce neutralizing antibody and cell-mediated immune responses against multiple coronavirus respiratory disease strains and variants/subvariants of SARS-CoV-2.

This is a randomized, open-label adjuvant dose-escalation study. The study will enroll healthy adults, aged 18 to 40 years of age, who had previously received two or more vaccinations with licensed COVID-19 vaccine(s), with the final dose administered a minimum of 6 months (24 weeks) prior to enrollment; have a negative PCR or rapid antigen SARS-CoV-2 test at screening; and have met all other eligibility criteria. Participants with a history of mild COVID-19 illness are eligible if they fully recovered a minimum of 6 months (24 weeks) prior to enrollment.

A total of 60 participants will be enrolled in the study. Study groups will be enrolled sequentially in an E6020 dose-escalating fashion starting with 20 participants to receive VBI-2901e with 1 µg of E6020 (Group G1), followed by 20 participants to receive VBI-2901e with 3 µg of E6020 (Group G2) and 20 participants to receive VBI-2901e with 10 µg E6020 (Group G3). Within each study group, participants will be randomized at a 1:1 ratio to receive one or two doses of VBI-2901e.

Group G1

* Subgroup G1-A: 10 participants to receive VBI-2901e at 5 µg with 1 µg E6020 per dose on Day 1.
* Subgroup G1-B: 10 participants to receive VBI-2901e at 5 µg with 1 µg E6020 per dose on Day 1 and Day 28.

Group G2

* Subgroup G2-A: 10 participants to receive VBI-2901e at 5 µg with 3 µg E6020 per dose on Day 1.
* Subgroup G2-B: 10 participants to receive VBI-2901e at 5 µg with 3 µg E6020 per dose on Day 1 and Day 28.

Group G3

* Subgroup G3-A: 10 participants to receive VBI-2901e at 5 µg with 10 µg E6020 per dose on Day 1.
* Subgroup G3-B: 10 participants to receive VBI-2901e at 5 µg with 10 µg E6020 per dose on Day 1 and Day 28.

The objective of the study is to select the optimal dose level of E6020 adjuvant (1, 3 or 10 μg) and number of doses (1 or 2 doses) of trivalent coronavirus vaccine candidate VBI-2901e in individuals who had been vaccinated against COVID-19 previously. To achieve this objective, the study will evaluate outcomes including safety and tolerability as well as antibody and T cell immune responses against the original SARS-CoV-2 ancestral strain, selected SARS-CoV-2 variants, SARS-CoV-1 and MERS-CoV.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject 18-40 years of age
2. Be willing and able to provide personally signed informed consent indicating understanding of the purpose, procedures required for the study and potential risks and benefits of the study, and be willing to participate in the study
3. Healthy participants with no chronic medical conditions at study enrollment and during the 6 months before enrollment. Participants with history of asymptomatic SARS-CoV-2 infection who tested positive by PCR or rapid antigen test or participants with history of having signs and symptoms mild COVID-19 illness (e.g., fever, cough, sore throat, malaise, headache, muscle pain, nausea, vomiting, diarrhea, loss of taste and smell) but who did not have shortness of breath, dyspnea, or abnormal chest imaging are eligible for the study if they fully recovered a minimum of 6 months before enrollment.
4. Meets reproductive inclusion criteria

   Female participant is eligible if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies:

   • is of childbearing potential and must have a negative pregnancy test prior to study vaccinations and agree to use an effective method of birth control as deemed appropriate by the investigator (e.g., hormonal contraceptive, barrier contraceptive with additional spermicide, or an intrauterine device) beginning >30 days prior to the first study vaccine administration and continuing for a minimum of 30 days after the last dose of study vaccine.

   OR

   • is not of childbearing potential, defined as postmenopausal (a minimum of 12 months with no menses without an alternative medical cause) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy).

   Male participant is eligible to participate if he agrees to the following requirements from the time of first study vaccination until at least 30 days after the last dose of study vaccine:
   * Be abstinent from heterosexual intercourse with a female of childbearing potential OR
   * Must agree to use a male condom. In addition to male condom use, an effective method of contraception may be considered in female partners of male participants AND
   * Must refrain from sperm donation
5. Have previously received 2 or more doses of a licensed COVID-19 vaccine(s) with the last dose administered a minimum of 6 months (24 weeks) prior to enrollment. Participants vaccinated with any of the vaccines approved by Health Canada for active immunization to prevent coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS- CoV-2) in individuals 18 years of age and older are eligible for the study. This includes the following COVID-19 vaccines: Moderna Spikevax®, Pfizer-BioNTech Comirnaty®, AstraZeneca Vaxzevria®, Janssen Jcovden® (Johnson & Johnson), Novavax Nuvaxovid® and Medicago Covifenz®. Participants who received one or more doses of VBI-2902a, VBI-2905a or any other COVID-19 vaccines that are either investigational or not approved by Health Canada are not eligible for the study.

Exclusion Criteria:

1. History of COVID-19 illness of moderate or greater severity, defined as one of the following:

   1. Moderate Illness: Individuals who show evidence of lower respiratory disease during clinical assessment or imaging and who have an oxygen saturation (SpO2) ≥94% on room air at sea level.
   2. Severe COVID-19 illness: Individuals who have SpO2 <94% on room air at sea level, a ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mm Hg, a respiratory rate >30 breaths/min, or lung infiltrates >50%.
   3. Critical COVID-19 illness: Individuals who have respiratory failure, septic shock, and/or multiple organ dysfunction.
2. Positive SARS-CoV-2 PCR or rapid antigen test at screening.
3. History of SARS or MERS.
4. Participant with a history of an underlying clinically significant acute or chronic medical condition or physical examination findings for which, in the opinion of the investigator, participation in the study would not be in the best interest of the participant (e.g., could compromise participant's wellbeing) or that could prevent, limit, or confound the protocol-specified assessments.
5. Individuals with medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
6. History of cancer requiring chemotherapy or radiation within 5 years.
7. Lack of participant's capacity (mental, social, behavioral), in the investigator's judgement, to provide informed consent for participation in the study.
8. Known or suspected impairment of immunological function, including but not limited to:

   1. autoimmune diseases (e.g., multiple sclerosis, type 1 diabetes, myasthenia gravis, Crohn's disease and other inflammatory bowel diseases, celiac disease, systemic lupus erythematosus, scleroderma, including diffuse systemic form and CREST syndrome, systemic sclerosis, dermatomyositis polymyositis, rheumatoid arthritis, juvenile idiopathic arthritis, autoimmune thyroiditis - including Hashimoto thyroiditis, Grave's or Basedow's disease, immune thrombocytopenic purpura, autoimmune hemolytic anemia, autoimmune hepatitis, psoriasis, vitiligo, vasculitis, Guillain- Barré syndrome, transverse myelitis, Addison's disease, Bell's palsy and alopecia areata) or abnormal or positive test result for any of the following tests at the study screening visit:

      * ANA (Antinuclear Antibody)
      * RF (Rheumatoid Factor)
      * tTG-IgA (Tissue Transglutaminase IgA Antibody)
      * CRP (C-Reactive Protein)
      * TGAB (Thyroglobulin Antibody)
   2. primary immunodeficiency disorders (e.g., common variable immune deficiency (CVID), defective phagocytic cell function and neutropenia syndromes, complement deficiency).
   3. secondary immunodeficiency disorders (e.g., Acquired Immunodeficiency Syndrome caused by Human Immunodeficiency Virus infection (HIV/AIDS), solid organ transplant, splenectomy)
9. History of allergic reactions or anaphylactic reaction to any vaccine component.
10. Known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV). Negative result of Anti-HIV, Anti-HCV and HBsAg testing at screening is required for eligibility.
11. Pregnant or breastfeeding or plans to conceive from 2 weeks before the study until the end of study.
12. Clinically significant abnormal physical examination, vital signs, or clinically significant abnormal values for hematology, serum chemistry or urinalysis at screening as determined by the investigator.
13. Any laboratory test abnormality that would be considered of Grade 1 severity or above (as per FDA grading guidelines) and is considered as clinically significant by the investigator. Grade 2 severity or above is exclusionary, regardless of clinical assessment.
14. Receipt of blood products or immunoglobulin within 90 days prior to enrollment or likely to require blood products during the study period.
15. Chronic administration (defined as more than 14 days in total) of immune-suppressive or other immune-modifying drug within 6 months prior to enrollment (for corticosteroids, this is defined as prednisone ≥20 mg/day or equivalent). Inhaled and topical steroids are allowed.
16. Immunization with attenuated vaccines (e.g., shingles) within 4 weeks prior to enrollment.
17. Immunization with inactivated vaccines (e.g., influenza) within 2 weeks prior to enrollment.
18. Participation in another clinical study within 30 days prior to enrollment. Participants who received one or more doses of VBI-2902a or VBI-2905a or other investigational COVID-19 vaccines are not eligible for the study.
19. Any skin abnormality or tattoo that would limit post-vaccination injection site assessment.
20. Family members of study site personnel.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Local reactions (solicited adverse events) within 7 days of study vaccination | Through 7 days after each vaccination
Systemic reactions (solicited adverse events) within 7 days of study vaccination | Through 7 days after each vaccination
Unsolicited adverse events within 28 days of study vaccination | Through 28 days after each vaccination
Serious adverse events within 28 days of study vaccination and end of study | Through end of study (approximately 1 year)
Medically-attended adverse events within 28 days of study vaccination and end of study | Through end of study (approximately 1 year)
Seroresponse rate against SARS-CoV-2 ancestral (Wuhan) strain | Study days 1, 28 and 56

SECONDARY OUTCOMES:
Seroresponse rate against SARS-CoV-2 variants of concern (Beta, Delta and Omicron) | Study days 1, 28 and 56
  Percent of participants with ≥ 4-fold rise in neutralizing antibody titer at 28 days after the first vaccination and, in participants receiving two doses, 28 days after the second vaccination, compared to baseline (Day 1)
Seroresponse rate against SARS-CoV-1 and MERS-CoV | Study days 1, 28 and 56
  Percent of participants with ≥ 4-fold rise in neutralizing antibody titer at 28 days after the first vaccination and, in participants receiving two doses, 28 days after the second vaccination, compared to baseline (Day 1)
Geometric mean titer (GMT) of SARS-CoV-2 neutralizing antibodies | Study days 1, 7, 28, 35, 56, 84, 168 and 336
  Geometric mean titer of SARS-CoV-2 neutralizing antibodies against SARS-CoV-2 ancestral (Wuhan) strain and variants of concern (Beta, Delta and Omicron), SARS-CoV-1 and MERS-CoV at days 1, 7, 28, 35, 56, 84, 168 and 336
Geometric mean fold rise (GMFR) in serum neutralizing antibody titer against SARS-CoV-2 ancestral (Wuhan) strain and variants of concern (Beta, Delta and Omicron), SARS-CoV-1 and MERS-CoV | Study days 1, 7, 28, 35, 56, 84, 168 and 336
  Geometric mean fold rise in serum neutralizing antibody titer against SARS-CoV-2 ancestral (Wuhan) strain and variants of concern (Beta, Delta and Omicron), SARS-CoV-1 and MERS-CoV at Days 7, 28, 35, 56, 84, 168 and 336 compared to baseline (Day 1)
GMT of serum IgG antibody to spike protein and receptor-binding-domain (RBD) against SARS-CoV-2 ancestral (Wuhan) strain, selected SARS-CoV-2 variants (Beta, Delta and Omicron), SARS-CoV-1 and MERS-CoV | Study days 1, 7, 28, 35, 56, 84, 168, and 336
  GMT of serum IgG antibody to spike protein and receptor-binding-domain (RBD) by enzyme-linked immunosorbent assay (ELISA) against SARS-CoV-2 ancestral (Wuhan) strain, selected SARS-CoV-2 variants (Beta, Delta and Omicron), SARS-CoV-1 and MERS-CoV at Days 1, 7, 28, 35, 56, 84, 168, and 336
GMFR in serum IgG antibody to spike protein and receptor-binding-domain (RBD) against SARS-CoV-2 ancestral (Wuhan) strain, selected SARS-CoV-2 variants (Beta, Delta and Omicron), SARS-CoV-1 and MERS-CoV | Study days 1, 7, 28, 35, 56, 84, 168, and 336
  GMFR in serum IgG antibody to spike protein and receptor-binding-domain (RBD) by enzyme-linked immunosorbent assay (ELISA) against SARS-CoV-2 ancestral (Wuhan) strain, selected SARS-CoV-2 variants (Beta, Delta and Omicron), SARS-CoV-1 and MERS-CoV at Days 7, 28, 35, 56, 84, 168, and 336 compared to baseline (Day 1)
Interferon-gamma-positive cells against spike protein from SARS-CoV-2 ancestral (Wuhan) strain, selected SARS-CoV-2 variants (Beta, Delta and Omicron), SARS-CoV-1 and MERS-CoV | Study days 1, 7, 28, 35, 56 and 84
  Geometric mean number of interferon-gamma-positive cells per million peripheral blood mononuclear cells (PBMCs) by ELISPOT using spike protein from SARS-CoV-2 ancestral (Wuhan) strain, selected SARS-CoV-2 variants (Beta, Delta and Omicron), SARS-CoV-1 and MERS-CoV at Days 1, 7, 28, 35, 56 and 84
Serum binding IgG subclasses | Study days 1, 7, 28, 35, 56 and 84
  Serum binding IgG subclasses as a marker of Th1 (IgG1 and IgG3) and Th2 (IgG4) dominated responses at Days 1, 7, 28, 35, 56 and 84

OTHER OUTCOMES:
GMT of neutralizing antibodies against potentially zoonotic beta-coronaviruses | Study days 1, 7, 28, 35, 56, 84, 168 and 336
  GMT of neutralizing antibodies against potentially zoonotic beta-coronaviruses (e.g., bat and pangolin isolates) at Days 1, 7, 28, 35, 56, 84, 168 and 336

CONTACTS AND LOCATIONS:
Overall Officials: William Cameron, MD, Principal Investigator — Ottawa Hospital
Locations (4):
- Canada (4):
  - Canadian Center for Vaccinology, Halifax, Nova Scotia
  - Red Maple Trials, Ottawa, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - CHU de Québec Université Laval, Québec, Quebec